CLINICAL TRIAL: NCT07275788
Title: An Exploratory Study of REGEND003 Kidney Progenitor Cells on Patients With Type 2 Diabetes Mellitus (T2DM) and Chronic Kidney Disease (CKD)
Brief Title: A Study of REGEND003 on Patients With Type 2 Diabetes Mellitus (T2DM) and Chronic Kidney Disease (CKD)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REGEND003-CKD-001
Record Dates: First submitted 2025-11-20; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM) and Chronic Kidney Disease (CKD)
Keywords: Type 2 Diabetes Mellitus; Chronic Kidney Disease; Cell Therapy; Kidney Progenitor Cells
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REGEND003 (Experimental): REGEND003 for dosage escalation
  Interventions: Biological: REGEND003
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: REGEND003 — REGEND003
  Arms: REGEND003
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
REGEND003, which consists of human kidney progenitor cells, demonstrates promising potential in repairing kidney injury. The purpose of this study is to assess the saftey and tolerability of REGEND003 on patients with Type 2 Diabetes Mellitus and Chronic Kidney Disease. It is an exploratory study with multi-centered, randomized, controlled, single-blinded, dose-escalated designs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 75 years at the time of signing the informed consent form;
* Diagnosed with Type 2 Diabetes Mellitus for at least 1 year;
* Diagnosed with Chronic Kidney Disease (CKD);
* Voluntarily sign the informed consent form, be able to cooperate in completing study-related procedures and examinations, capable of adequately recording or describing changes in their condition, and demonstrate strong compliance.

Exclusion Criteria:

* Females who are pregnant, nursing, or planning to be pregnant within a year after using this product (or males whose spouse planning to be pregnant);
* At the time of screening, subject who is positive in each of treponema pallidum antibody (TP-Ab), human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody test.

Hepatitis B virus carriers with stable current condition can be enrolled. Cured hepatitis C patients with negative result in HCV ribonucleic acid (RNA) test can be enrolled as well.

* Presence of a current or prior history of malignant tumor at screening (with the exception of those with disease-free survival for more than 2 years, or malignancies deemed to be of low aggressiveness as assessed by the investigator).
* Patients with Type 1 Diabetes Mellitus;
* Patients undergoing regular hemodialysis or peritoneal dialysis;
* Presence of severe acute complications of diabetes or CKD requiring hospitalization within 2 weeks prior to screening;
* Presence of more than one episode of hypoglycemic coma (blood glucose ≤3.9 mmol/L) within 1 month prior to screening;
* Patients intolerant to renal puncture/intrarenal injection procedures;
* Patients with diagnosis of acute kidney injury, congenital or hereditary kidney diseases, renal atrophy, or other renal conditions deemed ineligible by the investigator, as well as patients with a history of kidney transplantation at screening;
* Presence of severe systemic diseases within 6 months prior to screening and judged by the investigator as unsuitable for the study;
* Patients requiring long-term anticoagulant or antiplatelet therapy who, in the investigator's judgment, cannot discontinue medication 1 week prior to renal puncture/intrarenal injection procedures;
* Patients with suicidal risk, history of psychiatric disorders, or history of epilepsy at screening;
* Patients with severe arrhythmias or heart conduction disorders (degree II or above) in 12-lead ECG test at screening;
* Patients participated in other clinical trials with interventions within 1 month prior to screening;
* Subject with assessed survival time of less than 1 year by investigators at screening;
* Investigators, co-investigators, study coordinators, employees of participating investigators or research centers, or family members of the above individuals;
* Any condition that, in the investigator's judgment, may increase subject risk or interfere with the clinical trial.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event (AE) associated with the Cell Therapy | Within 24 weeks post-treatment
  The incidence and severity of adverse events will be evaluated.

SECONDARY OUTCOMES:
Complications associated with Intrarenal Injection | Within 24 weeks post-treatment
  The incidence will be evaluated.
Change from Baseline in Concentration of C-Reactive Protein | Within 24 weeks post-treatment
  C-Reactive Protein is a marker of inflammation in the body.
Change from Baseline in Glomerular Filtration Rate (GFR) | Within 24 weeks post-treatment
  GFR is a critical measurement of kidney function, reflecting how efficiently the kidneys filter blood
Change from Baseline in Concentration of Serum Creatinine | Within 24 weeks post-treatment
  A creatinine test is a measure of how well the kidneys are doing their job of filtering waste from the blood.
Change from Baseline in 24-Hour Urinary Protein Excretion | Within 24 weeks post-treatment
  A 24-hour urine protein test measures the amount of albumin (the most common protein filtered in the kidney) in the urine over 24 hours.
Change from Baseline in Urine Albumin-Creatinine Ratio (uACR) | Within 24 weeks post-treatment
  A urine albumin-creatinine ratio (uACR) is a urine (pee) test that help to understand the overall kidney health. A high uACR may be a sign of kidney disease.
Change from Baseline in Kidney Volume | Winthin 24 weeks post-treatment
  Kidney volume provides key insights in many clinical situations. Abnormal kidney volumes often signal problems.
Change from Baseline in Renal Cortical Thickness (RCT) | Within 24 weeks post-treatment
  RCT has also been used in the diagnosis of chronic kidney disease. With the progression of the disease, RCT decreases.
Changes from Baseline in the Outcomes from Kidney Disease Quality of Life (KDQOL) Survey | Within 24 weeks post-treatment
  The Kidney Disease Quality of Life (KDQOL) survey has long been used to assess the burden, symptoms/problems, and effects of kidney disease on a patient's quality of life. The minimal value is 0 and the maximal value is 100. A higher score means a better outcome.
Change from Baseline in Blood Pressure | Within 24 weeks post-treatment
  Both systolic and diastolic blood pressures are assessed.
Time from Injection to First Kidney Disease Progression (KDP) | Within 24 weekd post-treatment
  KDP is assessed by stage of disease, mortality and continous decreasing of GFR.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tongji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No